CLINICAL TRIAL: NCT05775484
Title: Exercise to Slow Cardiovascular Ageing Progression
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/2667
Record Dates: First submitted 2023-02-10; First posted 2023-03-20 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Ageing; Exercise; Cardiovascular
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- A: 1. Cardiovascular measurements Non-invasive brachial blood pressure machine Echocardiography
  2. Bio-specimen collection
  3. Six-minute walk test
  4. Musculoskeletal Analysis
  5. Cardiopulmonary exercise test
- B: 1. Cardiovascular measurements Non-invasive brachial blood pressure machine Echocardiography
  2. Bio-specimen collection
  3. Six-minute walk test
  4. Musculoskeletal Analysis
- C: 1. Cardiovascular measurements Non-invasive brachial blood pressure machine Echocardiography
  2. Bio-specimen collection
  3. Six-minute walk test
  4. Musculoskeletal Analysis
- D: 1. Cardiovascular measurements Non-invasive brachial blood pressure machine Echocardiography
  2. Bio-specimen collection
  3. Six-minute walk test (may require separate day visit to complete)
  4. Musculoskeletal Analysis
  5. Questionnaires

SUMMARY:
In ageing, deleterious alterations in cardiovascular (CV) structure and function increase risks of ageing-related cardiovascular disease (CVD). Investigators found that these CV alterations were associated with circulating serum metabolites, suggesting a metabolic basis to CV ageing. Investigators hypothesize that modification of these metabolites by intervention, such as exercise, may retard CV alterations and reduce CVD in ageing.

DETAILED DESCRIPTION:
Participants from each stratum will be randomized to receive either an exercise program intervention or no exercise. At the start and end of study, participants will undergo cardiovascular imaging and metabolic profiling. Investigators will determine if exercise can reverse high-risk metabolic profiles and improve cardiovascular structure and function.

Without clear mechanisms to explain cardiovascular ageing nor interventions known to retard cardiovascular ageing, our approach will provide much needed translational evidence to incorporate targeted interventions aimed at reducing cardiovascular disease risk in older populations.

ELIGIBILITY:
Inclusion Criteria:

* Age >=21 years old
* Outdoor ambulant

Exclusion Criteria:

* Wheelchair or bed-bound
* Dementia
* Residing in sheltered or nursing home
* Cancer
* Participation in ongoing clinical trials that involve interventional drugs or devices
* Aneurysms
* Acute infections (in the last six months)
* Uncontrolled thyrotoxicosis
* Neuromuscular, musculoskeletal or rheumatoid disorders that are exacerbated by exercise
* Uncontrolled asthma or chronic lung disease
* Restrictive lung disease

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruited through research studies and community studies.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolite profiles | 12 Months
  To measure changes in serum metabolite levels among participants pre and post exercise intervention.
Cardiovascular structure and function | 12 Months
  To measure changes in CV structure and function (diastolic function, arterial stiffness) among participants.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No